CLINICAL TRIAL: NCT04055883
Title: A Multicenter, Double-blind, Placebo-controlled, Stratified-randomized, Parallel, Therapeutic Exploratory Clinical Study to Evaluate the Efficacy and Safety of DA-1229 in Patients With Calcific Aortic Valve Disease
Brief Title: Clinical Study to Evaluate Efficacy and Safety of DA-1229 in Patients With CAVD
Acronym: DIP-CAVD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DA1229_CAVD_II
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Calcific Aortic Valve Disease
MeSH Terms: interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DA-1229 5mg (Experimental): Oral administration of DA-1229 5mg tablet once a day
  Interventions: Drug: DA-1229
- DA-1229 10mg (Experimental): Oral administration of DA-1229 10mg tablet once a day
  Interventions: Drug: DA-1229
- DA-1229 Placebo (Placebo Comparator): Oral administration of DA-1229 Placebo tablet once a day
  Interventions: Drug: DA-1229

INTERVENTIONS:
Drug: DA-1229 — All participants are administered one tablet per day for 96 weeks

SUMMARY:
This study will evaluate the efficacy and safety of DA-1229 in patients with calcific aortic valve disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects of ages in the range over 19
* The subjects whose echocardiography or heart CT result meets the criterion in the screening period or 4 weeks before screening visit

  * Criterion : 2.0m/s ≤ peak aortic-jet velocity < 4.0m/s or aortic valve calcium score ≥300AU
* The subjects completely understood the clinical trial through detailed explanation presented, determined to participate in the clinical trial spontaneously, and agreed to observe precautions suggested thereby through written consent

Exclusion Criteria:

* The cause of CAVD is niether degenerative nor bicuspid aortic valve
* The subjects who have other aortic valve disease as other clinically significant aortic insufficiency or mitral disease
* The subjects who had an aortic valve operation or are expected to need aortic valve operation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
aortic valve calcium volume change | 96 weeks
  aortic valve calcium volume change compared to baseline(mm^3)

SECONDARY OUTCOMES:
aortic valve calcium volume change | 48 weeks
  aortic valve calcium volume change compared to baseline(mm^3)
aortic valve calcium score change | 48 weeks, 96 weeks
  aortic valve calcium score change compared to baseline(AU)
aortic valve calcium volume change percent | 48 weeks, 96 weeks
  aortic valve calcium volume change percent compared to baseline(%)

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Seoul National University Bundang Hospital, Seongnam-si, Bundang-gu
  - Chonnam National University Hospital, Gwangju, Donggu
  - Gangnam Severance Hospital, Seoul, Gangnam-gu
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Kyeongpook National University Hospital, Daegu, Jung-gu
  - Chungnam National University Hospital, Daejeon, Jung-gu
  - Pusan National University Yangsan Hospital, Yangsan, Mulgeum-eup
  - Severance, Seoul, Seodaemun-gu
  - Asan Medical Center, Seoul, Songpa-gu

REFERENCES:
- [Derived] Song JK, Lee S, Kim YJ, Kim HK, Ha JW, Choi EY, Park SW, Park SJ, Park YH, Park JH, Yang DH, Kim KH, Yang DH, Han S, Chae SY, Lee JS, Song JM, Cho GY. Effect of Evogliptin on the Progression of Aortic Valvular Calcification. J Am Coll Cardiol. 2024 Sep 17;84(12):1064-1075. doi: 10.1016/j.jacc.2024.06.037. PMID 39260927